CLINICAL TRIAL: NCT04047160
Title: An Open-Label, Dose-Finding Study for the CBP / β-catenin Inhibitor OP-724 in Patients With Primary Biliary Cholangitis (Phase I)
Brief Title: Safety, Tolerability of OP-724 in Patients With Primary Biliary Cholangitis (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kiminori Kimura, MD (Other)
Collaborators: Ohara Pharmaceutical Co., Ltd. (Industry); Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Sponsor-Investigator, Kiminori Kimura, MD, Head, Department of Hepatology, Komagome Hospital
Organization: Komagome Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-724-P101; jRCT2031190073 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2019-07-30; First posted 2019-08-06 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Primary Biliary Cholangitis (PBC); Liver Cirrhosis, Biliary
Keywords: Primary Biliary Cholangitis (PBC); Liver Cirrhosis, Biliary; Cholangitis, Chronic Nonsuppurative Destructive; Liver Cirrhosis, Obstructive; Secondary Biliary Cholangitis; Primary Biliary Cirrhosis; Secondary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OP-724 (Experimental): Dose: 140, 280, 380 mg/m2/4 hrs
  Administration method:
  [Level 1] 140 mg/m2/4 hours [Level 2] 280 mg/m2/4 hours (starting dose) [Level 3] 380 mg/m2/4 hours Continuous intravenous administration will be done for 4 hours twice a week. This procedure will be as one cycle and 12 cycles (12 weeks in total) will be conducted. On 7 days prior to the first cycle administration, a dose scheduled in the first cycle will be administered with continuous intravenous for 4 hours and the safety and pharmacokinetics on the day of administration to the next day after administration will be evaluated.
  Interventions: Drug: OP-724

INTERVENTIONS:
Drug: OP-724 — Twice a week for 4 hours continuous intravenous administration of OP-724
  Other Names: CBP-beta-catenin inhibitor; PRI-724 (former name)

SUMMARY:
To evaluate the safety and pharmacokinetics of OP-724 and to determine the recommended dose of OP-724 against Primary Biliary Cholangitis patients.

DETAILED DESCRIPTION:
This trial is a phase I trial aimed at examining the safety and tolerability of OP-724 in patients with primary biliary cholangitis and determining the recommended dose.

The subjects are patients diagnosed with primary biliary cholangitis and diagnosed as progress of fibrosis (Scheuer stage III or higher) as a result of liver tissue examination. As a dosing schedule, OP-724 is intravenously administered twice a week (4 hours) for 12 weeks. However, once 7 days prior to the first cycle of administration, a dose scheduled for the first cycle will be administered once by continuous intravenous administration for 4 hours, and safety and pharmacokinetics will be evaluated on the day of administration to the next day after administration. The dose level shall be 3 doses (140 mg/m2/4hrs, 280 mg/m2/4hrs [starting dose], 380 mg/m2/4hrs), of which 2 doses shall be registered for up to 6 patients each. The safety and pharmacokinetic data after OP-724 administration will be decided comprehensively to determine the recommended dose in the next phase.

ELIGIBILITY:
Inclusion Criteria:

* (1) Of the confirmed patients * of primary biliary cholangitis, patients with progressive fibrosis (Scheuer classification stage III or higher) by liver biopsy.

  * The diagnosis of primary biliary cholangitis (PBC) is based on the diagnostic criteria (2015) of "Study and research on refractory liver and biliary diseases". That is, one that corresponds to any one of the following is diagnosed as PBC.
  1. Histologically, chronic non-suppurative destructive cholangitis (CNSDC) is found and the laboratory findings are consistent as PBC.
  2. A positive antimitochondrial antibody (AMA) with no histologic findings of CNSDC but showing a histology consistent with PBC.
  3. There is no experience of histologic search, but AMA is positive and it is considered as PBC from clinical image and course.
* (2) Patients with Performance Status 0 to 2.
* (3) Patients aged 20 years or over and under 75 when acquiring informed consent.
* (4) Regarding participation in this trial (including liver biopsy), patients who obtained informed consent by their own voluntary intention.

Exclusion Criteria:

* (1) Patients who have liver fibrosis other than primary biliary cholangitis or patients whose cause of liver fibrosis is unknown.
* (2) Patients with esophageal gastric varices determined to be treated by endoscopic examination at screening.
* (3) Patients with complication or previous history of primary liver cancer (excluding those who have had more than one year of hepatocarcinoma resection / radiofrequency ablation).
* (4) Merger of malignant tumor or past patients (within 3 years before screening). However, the following diseases are excluded: treated basal cell carcinoma, treated lung intraepithelial carcinoma, treated cervical carcinoma, or control superficial (not invasive) bladder carcinoma.
* (5) Patients who can not be denied hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), human T-cell leukemia virus 1 (HTLV-1) or syphilis.
* (6) Serum creatinine value: Patients with more than 1.5 times the upper limit of the facility reference value.
* (7) Patients with poor control of diabetes, hypertension or heart failure.
* (8) Patients with psychiatric diseases judged to have the potential to influence the implementation of clinical trials.
* (9) Patients who have severe allergy to or contrast media.
* (10) Patients whose dosage regimen was changed within 12 weeks prior to enrollment.
* (11) Patients who have history of drug or alcohol intoxication within 5 years before acquiring informed consent or who have history of drug or alcohol abuse within the past year.
* (12) Patients who participated in other clinical trials and clinical trials within 30 days prior to acquisition of consent, patients who used investigational drugs or investigational equipment.
* (13) Patients who received liver transplantation or other organ transplantation (including bone marrow transplantation) and patients who are difficult to intravenously administer.
* (14) Patients whose liver biopsy is expected to be difficult to perform.
* (15) Patients who are pregnant or nursing, or who are likely to become pregnant.
* (16) Male patients who do not obtain consent to contraception from the time of acquiring informed consent until the end of 12 weeks after the administration of investigational drug.
* (17) In addition, patients investigated by investigators or clinical trial doctors as judged unsuitable for this trial.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Occurrence Rate of Serious Adverse Events (Side Effects) | 28 days after the last administration of OP-724
  Occurrence Rate of Serious Adverse Events (Side Effects) whose causal relationship with the investigational drug can not be denied. The data will be aggregated by each adverse event and cohort.

SECONDARY OUTCOMES:
Expression Ratio of Adverse Events | 28 days after the last administration of OP-724
  The data will be aggregated by each adverse event and cohort.
Percentage of Occurrence of Side Effects | 28 days after the last administration of OP-724
  The data will be aggregated by each side effect and cohort.
Drug Concentration (OP-724 and C-82) in Plasma | A) Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours. / B) Continuous administration part: pre-dose and post-dose at 4 hours on Day 1 and 4 in Cycle 1, 5, 9 and 12 (each cycle is 7 days)
  The data will be aggregated by each cohort.
Parameters on Pharmacokinetics (OP-724 and C-82) : Maximum Plasma Concentration (Cmax) | A) Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours. / B) Continuous administration part: pre-dose and post-dose at 4 hours on Day 1 and 4 in Cycle 1, 5, 9 and 12 (each cycle is 7 days)
  The data will be aggregated by each cohort.
Parameters on Pharmacokinetics (OP-724 and C-82) : Area Under the Curve (AUC 0-24h) | A) Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours. / B) Continuous administration part: pre-dose and post-dose at 4 hours on Day 1 and 4 in Cycle 1, 5, 9 and 12 (each cycle is 7 days)
  The data will be aggregated by each cohort.
Liver Tissue Fibrotic Area Ratio by Liver Biopsy | 12 weeks after administration of OP-724
  Amount of change from baseline in liver tissue fibrotic area ratio by liver biopsy at 12 weeks after administration. The data will be aggregated by each cohort.
Liver Stiffness by Fibro Scan | 12 weeks after administration of OP-724
  Amount of change from baseline of liver stiffness by Fibro Scan at 12 weeks after administration. The data will be aggregated by each cohort.
Child-Pugh Score | 12 weeks after administration of OP-724
  Amount of change from baseline of Child-Pugh Score at 12 weeks after administration. Child Pugh score (scale range 5-15 points, the severity increases sequentially from 5 to 15 points) is obtained by adding the score for each parameter (hepatic encephalopathy, ascites, bilirubin, albumin, PT). Based on the total points score (Child-Pugh Score) of each diagnostic parameter shown above, the severity of the disease is classified into Grades A to C shown below. The data will be aggregated by each cohort and score.
  * Grade A: 5-6 points -> Compensated cirrhosis
  * Grade B: 7-9 points -> Decompensated cirrhosis
  * Grade C: 10-15 points -> Decompensated cirrhosis
MELD Score | 12 weeks after administration of OP-724
  Amount of change from baseline in MELD score at 12 weeks after administration. The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease and uses the subject's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. MELD is calculated according to the following formula:
  * MELD score = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43 The data will be aggregated by each cohort and score.
Modified Histological Activity Index (HAI) | 12 weeks after administration of OP-724
  Amount of change from baseline of modified Histological Activity Index (HAI) and classification of Nakanuma et al. by liver biopsy at 12 weeks after administration. The data will be aggregated by each cohort and index
Serum Alkaline Phosphatase (ALP) Level | 12 weeks after administration of OP-724
  Amount of change from baseline in serum ALP level at 12 weeks after administration. The data will be aggregated by each cohort and Child-Pugh score.
Serum Total Bilirubin Value | 12 weeks after administration of OP-724
  Amount of change from baseline in serum total bilirubin value at 12 weeks after administration. The data will be aggregated by each cohort and Child-Pugh score.
Enhanced Liver Fibrosis Panel (ELF) Score | 12 weeks after administration of OP-724
  Amount of change from baseline of ELF score at 12 weeks after administration. Observation items: hyaluronic acid, procollagen III peptide, TIMP-1
  * ELF score = 2.278 + 0.851 ln (hyaluronic acid) + 0.75 ln (P3 NP) + ln (TIMP). The data will be aggregated by each cohort and score.

OTHER OUTCOMES:
Effectiveness: Serum Fibrosis Marker Level | 12 weeks after administration of OP-724
  Amount of change from baseline in serum fibrosis marker level at 12 weeks after administration. The data will be aggregated by each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Kiminori Kimura, MD, Principal Investigator — Tokyo Metropolitan Komagome Hospital
Locations (2):
- Japan (2):
  - Tokyo Metropolitan Komagome Hospital, Bunkyō-Ku, Tokyo
  - Kyushu University Hospital, Fukuoka

REFERENCES:
- [Derived] Kimura M, Ogawa E, Harada K, Imamura J, Saio M, Ikura Y, Yatsuhashi H, Murata K, Miura K, Ieiri I, Tanaka A, Kimura K. Feasibility, safety and tolerability of the CREB-binding protein/beta-catenin inhibitor OP-724 in patients with advanced primary biliary cholangitis: an investigator-initiated, open-label, non-randomised, two-centre, phase 1 study. BMJ Open Gastroenterol. 2022 Nov;9(1):e001001. doi: 10.1136/bmjgast-2022-001001. PMID 36442892